CLINICAL TRIAL: NCT01349231
Title: Ketamine Infusion for Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901004660
Record Dates: First submitted 2011-04-09; First posted 2011-05-06 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Obsessive-compulsive Disorder
Keywords: obsessive-compulsive disorder; ketamine; glutamate
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine (Experimental): Ketamine will be given at a dose of 0.5mg/kg over 40 minutes. This dose is identical to that used in previous anti-depressant studies of ketamine.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — Ketamine (a single 0.5mg intravenously over 40 minutes).

SUMMARY:
Roughly one-third of patients with obsessive-compulsive disorder (OCD) do not experience significant clinical benefit from first-line interventions such as pharmacotherapy with selective serotonin reuptake inhibitors (SSRI) or cognitive behavioral therapy (CBT). Furthermore, OCD patients typically experience the full treatment benefits of first-line interventions only after a time-lag of two to three months. Inadequate symptom relief and delay of symptom relief from first-line treatments are sources of substantial morbidity and decreased quality of life in OCD patients. Converging lines of evidence from neuroimaging, genetic and pharmacological studies support the importance of glutamate abnormalities in the pathogenesis of OCD.

The investigators are conducting an open, uncontrolled study of ketamine in treatment-refractory OCD. Ketamine is a potent antagonist of the N-methyl-D-aspartate (NMDA) receptor and has been demonstrated to have rapid anti-depressant effects in patients with Major Depressive Disorder. The investigators have additionally provided evidence for rapid improvement of comorbid OCD and trichotillomania after ketamine infusion in a depressed woman.

Failure of symptom relief and delay of symptom relief from first-line treatments are a source of substantial morbidity and decreased quality of life in OCD patients. Ketamine represents the possibility to provide rapid symptom relief to OCD patients and may provide the mechanism for future drug development to treat OCD more rapidly and effectively.

DETAILED DESCRIPTION:
Roughly one-third of patients with obsessive-compulsive disorder (OCD) fail to experience significant clinical benefit from first-line interventions such as pharmacotherapy with selective serotonin reuptake inhibitors (SSRI) or cognitive behavioral therapy (CBT). Antipsychotic augmentation is the only pharmacological strategy for treatment-refractory OCD with demonstrated efficacy in multiple double-blind trials (2). Antipsychotic augmentation only benefits around 1 in 3 treatment-refractory OCD. Furthermore, OCD patients typically experience the full treatment benefits of first-line interventions only after a time-lag of two to three months. Failure of symptom relief and delay of symptom relief from first-line treatments are sources of substantial morbidity and decreased quality of life in OCD patients.

Converging lines of evidence from neuroimaging, genetic and pharmacological studies support the importance of glutamate abnormalities in the pathogenesis of OCD. In Magnetic Resonance Spectroscopy studies elevated concentrations of glutamate and related compounds have been demonstrated in the caudate nucleus and orbitofrontal cortex of OCD patients compared to normal controls. In genetic studies, single nucleotide polymorphisms within the glutamate transporter gene SLC1A1 have been associated with the diagnosis of OCD. Open-label, pharmacological treatment studies have suggested that glutamate modulating agents such as riluzole, n-acetylcysteine and memantine may be effective in the treatment of OCD.

Ketamine is a potent antagonist of the N-methyl-D-aspartate (NMDA) receptor, a major type of glutamate receptor in the brain. In a placebo-controlled study completed at Yale a single dose of ketamine (0.5 mg/kg, intravenously) had rapid antidepressant effects in depressed patients. In these subjects ketamine infusion produced mild psychotomimetic symptoms and euphoria that dissipated within 120 minutes, while the antidepressant effects of ketamine infusion emerged over the first 180 minutes and persisted over 72 hours. Fifty percent of depressed patients receiving ketamine were treatment responders at Day 3 compared to 12.5% in the placebo infusion group. These results have been replicated in a recent double-blind study performed at NIMH and a third unpublished study conducted by members of our group at Yale.

Our goal is to conduct an open-label study in treatment-refractory OCD to determine if ketamine may be an effective acute anti-obsessional agent.

ELIGIBILITY:
Inclusion Criteria:

1. Adult between the ages of 18 and 65 years.
2. Meet DSM IV criteria for obsessive-compulsive disorder by structured clinical interview (SCID) and have a Y-BOCS score >24.
3. Have treatment-refractory OCD. Have Y-BOCS>24 despite two SSRI trials of adequate dose and duration and been offered prior CBT treatment.
4. Stable psychiatric medications. Subjects must have had stable doses of all psychiatric medications for the month prior to treatment and have been on stable doses of SSRI and clomipramine for at least 2 months prior to study enrollment.
5. Medically and neurologically healthy.
6. Able to provide written informed consent according to the Yale HIC guidelines.

Exclusion Criteria:

1. Lifetime history of substance dependence (other than nicotine and caffeine)
2. Suicide attempt or suicidal ideation requiring psychiatric hospitalization in the previous 6 months
3. Being Pregnant
4. Known hypersensitivity to ketamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center/ YNHH, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Niciu MJ, Grunschel BD, Corlett PR, Pittenger C, Bloch MH. Two cases of delayed-onset suicidal ideation, dysphoria and anxiety after ketamine infusion in patients with obsessive-compulsive disorder and a history of major depressive disorder. J Psychopharmacol. 2013 Jul;27(7):651-4. doi: 10.1177/0269881113486718. Epub 2013 May 15. PMID 23676198
- See also: Yale OCD Research Clinic — http://psychiatry.yale.edu/research/programs/clinical_people/ocd.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) [Mean (Standard Deviation); unit: units on a scale] — The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) assesses obsessive and compulsive symptom severity. Obsessions are rated on a scale from 0-20 and compulsions are rated on a scale of 0-20 for a total scale of 0-40. Scores on the obsessions scale and scores on the compulsions scale are summed to obtain the total score. Lower values represent better outcomes.
  units on a scale | 32.9 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: OCD Severity
Description: We will examine change from baseline in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) ratings of OCD severity at 1 day following infusion. The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) assesses obsessive and compulsive symptom severity. Obsessions are rated on a scale from 0-20 and compulsions are rated on a scale of 0-20, for a total scale of 0-40. Scores on the obsessions scale and scores on the compulsions scale are summed to obtain the total score. The higher the score, the more severe the OCD.
Time Frame: Baseline and 1 day after ketamine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
units on a scale | -2.7 (1.11)

2. Primary Outcome: OCD Severity
Description: We will examine change from baseline in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) ratings of OCD severity at 2 days following infusion. The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) assesses obsessive and compulsive symptom severity. Obsessions are rated on a scale from 0-20 and compulsions are rated on a scale of 0-20, for a total scale of 0-40. Scores on the obsessions scale and scores on the compulsions scale are summed to obtain the total score. The higher the score, the more severe the OCD.
Time Frame: Baseline and 2 days following infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
units on a scale | -3.6 (1.19)

3. Primary Outcome: OCD Severity
Description: We will examine change from baseline in the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) ratings of OCD severity at 3 days following infusion. The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) assesses obsessive and compulsive symptom severity. Obsessions are rated on a scale from 0-20 and compulsions are rated on a scale of 0-20, for a total scale of 0-40. Scores on the obsessions scale and scores on the compulsions scale are summed to obtain the total score. The higher the score, the more severe the OCD.
Time Frame: Baseline and 3 days following infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
units on a scale | -2.9 (0.91)

4. Secondary Outcome: Depression Symptoms
Description: We will examine change from baseline in Hamilton Rating Scale for Depression (HRDS) ratings of depression severity at day 1-3 following a single ketamine infusion. The HRDS assesses severity of, and change in, depressive symptoms. The HRDS is a 21 item scale with scores ranging from 0-66. The higher the score, the more severe the depression.
Time Frame: Baseline, Day 1, Day 2, and Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 10
units on a scale
  HRDS change from Baseline to Day 1 | -6.57 (1.69)
  HRDS change from Baseline to Day 2 | -7.29 (2.89)
  HRDS change from Baseline to Day 3 | -5.14 (2.48)

ADVERSE EVENTS:
Arm/Group | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=10)
Transient increase in systolic blood pressure (General disorders) | 1 — 30% above baseline, maximum 160/80, which lasted 10 min
Dysphoria (Psychiatric disorders) | 2
Dissociative symptoms (Psychiatric disorders) | 5 — Gaps in memory(n=3), sensory distortions (i.e., perioral perasthesias, n=2), a feeling that time was moving in slow motion (n=2), and disconnected feeling from reality (n=1). No subjects reported any dissociative symptoms beyond the 1-hour time point
Anxiety (Psychiatric disorders) | 2
Passive suicidal ideation (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes